CLINICAL TRIAL: NCT05188313
Title: The Efficacy of the Addition of TRAstuzumab and Pertuzumab to Neoadjuvant Chemoradiation: a Randomized Multi-center Study in Resectable HER2 Overexpressing Adenocarcinoma of the Esophagus or Gastroesophageal Junction. The TRAP-2 Study
Brief Title: TRAstuzumab and Pertuzumab for HER2+ Resectable Oesophageal Cancer
Acronym: TRAP-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, Prof. dr. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79276.018.21
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Esophageal Cancer; Esophageal Adenocarcinoma
Keywords: HER2
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus | interventions — Trastuzumab; pertuzumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemoradiation according to the CROSS regimen (Active Comparator): Paclitaxel 50 mg/m2 and carboplatin AUC = 2 will be given by intravenous infusion on days 1, 8, 15, 22 and 29.
  A total dose of 41.4 Gy will be given in 23 fractions of 1.8 Gy, 5 fractions per week, starting the first day of the first cycle of chemotherapy.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Chemoradiation according to the CROSS regimen combined with trastuzumab and pertuzumab (Experimental): Paclitaxel 50 mg/m2 and carboplatin AUC = 2 will be given by intravenous infusion on days 1, 8, 15, 22 and 29.
  A total dose of 41.4 Gy will be given in 23 fractions of 1.8 Gy, 5 fractions per week, starting the first day of the first cycle of chemotherapy.
  Pertuzumab will be administered intravenously first, on Day 1, 22, 43, 64, and 85 using a fixed dose of 840 mg.
  Trastuzumab will be administered intravenously on Day 1 of each treatment cycle, using an initial dose of 4 mg/kg on day 1, followed by doses of 2 mg/kg weekly up to week 6. From week 7 onwards trastuzumab will be administered at a dose of 6 mg/kg, every three weeks.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Trastuzumab — Intravenous administration of study drug
  Arms: Chemoradiation according to the CROSS regimen combined with trastuzumab and pertuzumab
Drug: Pertuzumab — Intravenous administration of study drug
  Arms: Chemoradiation according to the CROSS regimen combined with trastuzumab and pertuzumab
Drug: Paclitaxel — Intravenous administration of study drug
Drug: Carboplatin — Intravenous administration of study drug

SUMMARY:
Despite treatment according to the CROSS-regimen, median overall survival is less than four years (2.3 QALYs). The burden of disease is within the highest category (0.71 to 1.0). Also, no targeted treatment options are currently available, hampering personalized treatment for this patient population. TRAP-2 aims to address these needs by investigating whether addition of trastuzumab and pertuzumab to standard of care improves survival of patients with resectable HER2 positive esophageal adenocarcinoma (HER2+ EAC). Patients with HER2+ EAC will be randomised to neoadjuvant chemoradiation according to the CROSS regimen or CROSS + TRAstuzumab and Pertuzumab. Primary outcome is overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the esophagus or gastroesophageal junction, T1N+M0; or T2-T4a N0 or N+ M0).
* HER2-positive tumor defined as either IHC 3+ or IHC 2+, the latter in combination with ISH+, as assessed by the local laboratory on a primary tumor biopsy. HER2 status needs to be confirmed by the central laboratory, but does not affect start of treatment.
* Surgical resectability, as determined during multidisciplinary meeting. Tumors that cannot be passed with an endoscope for endoscopic ultrasound are eligible if all other criteria are fulfilled.
* If the tumor extends below the gastroesophageal (GE) junction into the proximal stomach, the bulk of the tumor must involve the esophagus or GE junction.
* Age ≥ 18.
* ECOG performance status 0 or 1 (cf. Appendix A).
* Adequate hematological, renal and hepatic functions defined as:

  * Neutrophils ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 5.6 mmol
  * Total bilirubin ≤ 1.5 x upper normal limit
  * Creatinine clearance (Cockroft) > 60 ml/min
* Adequate left ventricular ejection fraction defined as an LVEF of ≥55% determined by transthoracic echocardiography or MUGA.
* Written, voluntary informed consent
* Patients must be accessible to follow up and management in the treatment center

Exclusion Criteria:

* T1N0 tumors or in situ carcinoma.
* Past (within 5 years) or current history of malignancy other than entry diagnosis which has a worse expected prognosis than the current esophageal cancer.
* Previous chemotherapy, radiotherapy, treatment with an anti-HER2 antibody or with small molecule HER2 inhibitors for esophageal cancer or for any other cancer within 6 months of diagnosis of esophageal cancer.
* Previous radiation to the mediastinum precluding full dose radiation of the currently present esophageal tumor.
* Invasion of the tracheobronchial tree or presence of tracheoesophageal fistula.
* Pregnancy (positive serum pregnancy test), planning to become pregnant, and lactation.
* Not willing to use highly effective methods of contraception (per institutional standard) during treatment (male or female) and for 6 months after the end of treatment.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) precluding major surgery.
* Pulmonary fibrosis and/or severely impaired lung function (FEV1 < 1,5L) precluding major surgery.
* Serious underlying medical condition which would impair the ability of the patient to receive the planned treatment, including prior allergic reactions to drugs containing Cremophor, such as teniposide or cyclosporine.
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Inadequate caloric- and/or fluid intake despite consultation of a dietician and/or tube feeding.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Active infection requiring systemic therapy which has not resolved 3 days (simple infection such as cystitis) to 7 days (severe infection such as pyelonephritis) prior to the first dose of trial treatment.
* Evidence of acute or chronic infection with hepatitis B, C or HIV.
* History of prior allogeneic stem cell or solid organ transplantation.
* Pre-existing motor or sensory neurotoxicity greater than or equal to CTC AE grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2037-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5.5. years (maximum follow-up time)
  Overall survival will be calculated from the date of randomization to death.

SECONDARY OUTCOMES:
Progression free survival | 5.5. years (maximum follow-up time)
  Progression free survival will be calculated from the date of randomization to death or progression.
Adverse events | 15 weeks (duration of neoadjuvant treatment)
  Treatment toxicity according
Surgical complications | 30 days after surgery
  Surgical complications according to Clavien Dindo
Left Ventricular Systolic Dysfunction | 5.5. years
  ≥ 10 percentage points decrease from baseline to an absolute value < 50%
General quality of life | 5.5. years
  Quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided